CLINICAL TRIAL: NCT01180816
Title: Phase I Trial of Super-Selective Intraarterial Cerebral Infusion of Temozolomide (Temodar) for Treatment of Newly Diagnosed Glioblastoma Multiforme and Anaplastic Astrocytoma
Brief Title: Super-Selective Intraarterial Cerebral Infusion Of Temozolomide (Temodar) For Treatment Of Newly Diagnosed GBM And AA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other); Hofstra North Shore (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor, Feinstein Institute for Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-292A
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: GBM; AA; AO; Brain; Tumors; Malignant; Glioblastoma; Multiforme; Anaplastic; Astrocytoma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide (Temodar) (Experimental)
  Interventions: Drug: Super-Selective Intraarterial Intracranial Infusion of Temozolomide

INTERVENTIONS:
Drug: Super-Selective Intraarterial Intracranial Infusion of Temozolomide — A single dose of Intraarterial Mannitol to open the blood brain barrier followed by Intra-arterial Temozolomide single dose (starting at 75mg/m2 and up to 250mg/m2)

SUMMARY:
The high-grade malignant brain tumors, glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA), comprise the majority of all primary brain tumors in adults. This group of tumors also exhibits the most aggressive behavior, resulting in median overall survival durations of only 9-12 months for GBM, and 3-4 years for AA. Initial therapy has consisted of surgical resection, external beam radiation or both. More recently, a Phase 3 clinical published by Stupp et al in 2005 showed a benefit for using radiotherapy plus concomitant and adjuvant Temozolomide. Still, all patients experience a recurrence after first-line therapy, so improvements in both first-line and salvage therapy are critical to enhancing quality-of-life and prolonging survival. It is unknown if currently used intravenous (IV) therapies even cross the blood brain barrier (BBB). Superselective Intra-arterial Cerebral Infusion (SIACI) is a technique that can effectively increase the concentration of drug delivered to the brain while sparing the body of systemic side effects. One currently used drug called Temozolomide (Temodar) has been shown to be active in human brain tumors but its actual central nervous system (CNS) penetration is unknown. This phase I clinical research trial will test the hypothesis that following the standard 42 day Temozolomide/radiotherapy regimen, Temozolomide can be safely used by direct intracranial superselective intra-arterial cerebral infusion (SIACI) up to a dose of 250mg/m2, followed by the standard maintenance cycle of temozolomide to ultimately enhance survival of patients with newly diagnosed GBM/AA. The investigators will determine the toxicity profile and maximum tolerated dose (MTD) of SIACI Temozolomide. The investigators expect that this project will provide important information regarding the utility of SIACI Temozolomide therapy for malignant gliomas, and may alter the way these drugs are delivered to our patients in the near future.

DETAILED DESCRIPTION:
The current standard of care for newly diagnosed GBM is radiation therapy plus concomitant oral Temozolomide of doses of 75mg/m2 up to 150mg/m2. Because of the blood brain barrier (BBB) where drugs do not penetrate the blood vessel walls well to get into the brain, no one knows for sure if these oral drugs actually get into the brain after infusion. Previous studies have shown that intra-carotid artery (intra-arterial) delivery is superior to standard intravenous or oral delivery for increasing the penetration of drug to the brain. Previous techniques using intra arterial (intracarotid) infusion still were non-selective as drug delivery still went to all blood vessels in the brain, so patients still had significant adverse events, such as blindness. Newer techniques in interventional neuroradiology have allowed for a more selective delivery of catheters into the arterial tree where chemotherapies can be delivered without the risk of adverse affects such as blindness. Therefore, this trial will ask one simple question: Is it safe to deliver a dose of Temozolomide intraarterially using these super selective delivery techniques in addition to the standard oral route of administration? This should not only increase the amount of drug that gets to the tumor but also spare the patient many of the adverse effects from a less selective delivery. Prior to this single dose of intra-arterial Temozolomide, the patient will also receive a dose of mannitol that will increase the permeability of the blood brain barrier to improve delivery of the agent to the brain. After this single dose of mannitol and Temozolomide, the patient will be evaluated for 4 weeks to assess for toxicity. If there is no toxicity at this point, then the patient will proceed with oral maintenance Temozolomide chemotherapy. In summary, this is a Phase I trial that is designed to test the safety of a single dose of intra-arterial delivery of Temozolomide immediately following 42 days of radiotherapy/oral temozolomide and prior to starting oral maintenance Temozolomide.

To summarize:

Current Standard of Care Therapy:

Days 1-42: Adjuvant dose of Temozolomide 75mg/m2 for 42 days concomitant with focal radiotherapy Day 42: 4 week rest period Day 70: Maintenance dose of Temozolomide 150mg/m2 once daily for Days 1-5 of a 28 day cycle for 6 cycles

Experimental portion of this proposal:

Days 1-42: Adjuvant dose of Temozolomide 75mg/m2 for 42 days concomitant with focal radiotherapy Day 42: Single Intra-arterial Mannitol to increase the permeability of the blood brain barrier followed by Intra-arterial Temozolomide single dose (starting at 75mg/m2 and up to 250mg/m2) followed by 4 week rest period Day 70: Maintenance dose of Temozolomide 150mg/m2 once daily for Days 1-5 of a 28 day cycle for 6 cycles

Therefore the experimental aspects of this treatment plan will include:

1. On day 42, subjects will first be treated with Mannitol prior to chemotherapy infusion (Mannitol 25%; 3-10 mLs for 30seconds) in order to disrupt the blood brain barrier. This technique has been used in several thousand patients in previous studies for the intraarterial (IA) delivery of chemotherapy for malignant glioma.
2. Following the addition of mannitol, the investigators will deliver a single SIACI dose of Temozolomide for patients with high-grade glioma. After a one-cycle observation period to assess for toxicity from the IA infusion, the subject will receive the standard oral maintenance regimen of Temozolomide chemotherapy. The Intra-Arterial Infusion Procedure will be done under general anesthesia and standard monitoring will occur.

The dose escalation algorithm is as follows: The investigators will use a single intracranial superselective intra-arterial infusion of Temozolomide, starting at a dose of 75mg/m2 in the first three patients. Assuming no dose limiting toxicity during the next 28 days after the infusion, the patient will then begin standard maintenance oral Temozolomide chemotherapy regimen. The doses will be escalated from 75 to 100, to 150, 200, and finally 250mg/m2 in this Phase I trial.

Most patients with GBM are also monitored every two months with serial history, neurological and physical examinations together with serial blood counts, prothrombin time (PT), partial thromboplastin time (PTT) and chemistries. In addition, most patients with GBM have an MRI performed every two cycles or approximately every two months to assess for tumor progression. .

Since this is a Phase I trial, response is not a primary endpoint. However, the investigators will evaluate response to the one time IA Temozolomide therapy with a MRI with the injection of contrast approximately 4 weeks after infusion. Follow-up of all patients in the trial after the IA Temozolomide therapy will continue until disease progression or death. Survival will be measured from the time of the dose of IA Temozolomide®. The investigators expect patients in the trial to be monitored for 12 months.

ELIGIBILITY:
Criteria for Inclusion:

* Male or female patients of ≥18 years of age.
* Patients with a documented histologic diagnosis of newly diagnosed or glioblastoma multiforme (GBM), anaplastic astrocytoma (AA) or anaplastic mixed oligoastrocytoma (AOA).
* Patients must have at least one confirmed and evaluable tumor site.∗

  *A confirmed tumor site is one in which is biopsy-proven. NOTE: Radiographic procedures (e.g., Gad-enhanced MRI or CT scans) documenting existing lesions must have been performed within three weeks of treatment on this research study.
* Patients must have a Karnofsky performance status ≥60% (or the equivalent ECOG level of 0-2) and an expected survival of ≥ three months.
* No other chemotherapy for two weeks prior to treatment under this research protocol
* Patients must have adequate hematologic reserve with WBC≥3000mm3, absolute neutrophils ≥1500mm3 and platelets ≥100,000 mm3. Patients who are on Coumadin must have a platelet count of ≥150,000 mm3
* Pre-enrollment chemistry parameters must show: bilirubin<1.5X the institutional upper limit of normal (IUNL); AST or ALT<2.5X IUNL and creatinine<1.5X IUNL.
* Pre-enrollment coagulation parameters (PT and PTT) must be ≤1.5X the IUNL.
* Concomitant Medications:
* Growth factor(s): Must not have received within 1 week of entry onto this study.
* Steroids: Systemic corticosteroid therapy is permissible in patients with CNS tumors for treatment of increased intracranial pressure or symptomatic tumor edema. Patients with CNS tumors who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to study entry.
* Patients must agree to use a medically effective method of contraception during and for a period of three months after the treatment period. A pregnancy test will be performed on each premenopausal female of childbearing potential immediately prior to entry into the research study.
* Patients on steroids must receive prophylaxis for PCP pneumonia with Bactrim, unless they have a history of allergy to sulfa drugs.
* Patients must be able to understand and give written informed consent. Informed consent must be obtained at the time of patient screening.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Subjects who decline birth control. Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this research trial and will be advised that they must use effective contraception during and for a period of three months after the treatment period.
* Patients with significant intercurrent medical or psychiatric conditions that would place them at increased risk or affect their ability to receive or comply with treatment or post-treatment clinical monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2017-12 (Actual); Study Completion 2020-08-11 (Actual)

PRIMARY OUTCOMES:
Determine the safety of superselective intra-arterial cerebral infusion of Temozolomide up to a dose of 250 mg/m2 IA. | 2 years

SECONDARY OUTCOMES:
Composite overall response rate. | 2 years
Six-month progression-free survival (PFS) and overall survival (OS) | throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States